CLINICAL TRIAL: NCT02044263
Title: Cognitive Behavior Therapy for Insomnia Delivered by a Therapist or on the Internet: a Randomized Controlled Noninferiority Trial
Brief Title: Cognitive Behavior Therapy for Insomnia Delivered by a Therapist or on the Internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1836
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Insomnia
Keywords: Cognitive therapy; Behavior therapy; Waiting lists; Therapy, computer-assisted; Internet
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet CBT-i (Experimental): Participants will be instructed on the use of the internet CBT-i (SHUTi) intervention site, then use the program for six weeks.
  Interventions: Behavioral: Internet CBT-i SHUTi
- face-to-face CBT-i (Active Comparator): 4 to 8 sessions of face-to-face CBT-i treatment with one of three clinicians (experienced CBT-i psychiatrists)
  Interventions: Behavioral: face-to-face CBT-i

INTERVENTIONS:
Behavioral: Internet CBT-i SHUTi — Computer program SHUTi is based on the same theoretical model of insomnia and involves the same interventions as ordinary CBT-I: a structured treatment focusing on education, behaviors and cognitions. Specifically, CBT-I usually consists of one or more of the following: psychoeducation about sleep, sleep restriction therapy, stimulus control, relaxation techniques, and challenging beliefs and perception of sleep.
  Arms: Internet CBT-i
Behavioral: face-to-face CBT-i
  Arms: face-to-face CBT-i

SUMMARY:
Background: Insomnia is a highly prevalent and disabling disorder where Cognitive Behavior Therapy for Insomnia (CBT-I) is established as the best available treatment. Still, only a negligible number of patients with insomnia receive this treatment. One potential way of improving the dissemination of CBT-I is by using online adaptations of CBT-I. This is a new method for delivering CBT-I and it is not known how effective online treatment is compared to face-to-face CBT-I. This trial's purpose is to compare face-to-face CBT-I with online CBT-I. Because of the great advantage of online treatment in both availability and cost, the trial is designed as a noninferiority trial.

Aim: To test if online CBT-I is noninferior in reducing insomnia complaints compared with CBT-I as delivered face-to-face by a therapist.

ELIGIBILITY:
Inclusion Criteria:

* meeting the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnostic criteria for insomnia disorder

Exclusion Criteria:

* a condition that renders the patient incapable of understanding the treatment (e.g. actively psychotic, mental retardation, dementia or others
* an ongoing substance abuse problem
* other organic sleep disturbances or circadian sleep disturbance
* an ongoing medical condition where treatment of insomnia is not indicated (e.g. an attack phase of multiple sclerosis)
* working night shifts and being unable to discontinue this work pattern
* not being sufficiently fluent in Norwegian to understand the assessments or treatment
* not having the necessary computer skills needed to log on to the web based program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
insomnia severity | 6 months
  as assessed by Insomnia Severity Index (Morin ea 2011 Sleep 34(5):601-8)
insomnia severity | 8 weeks
  as assessed by Insomnia Severity Index (Morin ea 2011 Sleep 34(5):601-8)

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Kallestad, PhD PsyD, Principal Investigator — St. Olavs Hospital
Locations (1):
- Sleep Clinic, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] H Kallestad, K Langsrud, Ø Vedaa, T Stiles, D Vethe, S Lydersen, L Ritterband, G Morken, B Sivertsen. A Randomized Noninferiority Trial Comparing Cognitive Behavior Therapy For Insomnia (cbt-i) Delivered By A Therapist Or Via A Fully Automated Online Treatment Program. Sleep, Volume 41, Issue suppl_1, April 2018, Page A142 https://doi.org/10.1093/sleep/zsy061.370
- [Derived] Kallestad H, Scott J, Vedaa O, Lydersen S, Vethe D, Morken G, Stiles TC, Sivertsen B, Langsrud K. Mode of delivery of Cognitive Behavioral Therapy for Insomnia: a randomized controlled non-inferiority trial of digital and face-to-face therapy. Sleep. 2021 Dec 10;44(12):zsab185. doi: 10.1093/sleep/zsab185. PMID 34291808